CLINICAL TRIAL: NCT05090787
Title: Clinical Investigation of the TECNIS 1-Piece Intraocular Lens
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Business Decision
Sponsor: Johnson & Johnson Surgical Vision, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: CHVL-101-UACC
Record Dates: First submitted 2021-10-12; First posted 2021-10-25 (Actual); Last update posted 2024-02-06 (Actual); Status verified 2024-01

CONDITIONS: Cataract
MeSH Terms: conditions — Cataract

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (2):
- Investigational Device (Experimental): Investigational mDCB00
  Interventions: Device: Investigational mDCB00
- Control Device (Active Comparator): Control DCB00
  Interventions: Device: Control DCB00

INTERVENTIONS:
Device: Investigational mDCB00 — Investigational intraocular lens replaces the natural lens removed during cataract surgery in both eyes.
  Arms: Investigational Device
Device: Control DCB00 — Control intraocular lens replaces the natural lens removed during cataract surgery in both eyes
  Arms: Control Device

SUMMARY:
This study is a 6-month, prospective, comparative, multicenter, bilateral, parallel group, randomized (2:1), subject/evaluator masked clinical investigation of the investigational mDCB00 IOL as compared to the DCB00 IOL.

The study will be conducted at up to 8 sites in countries where both the investigational and control lenses are approved for market and/or for evaluation in a clinical study and will include a total of up to 200 subjects. Subjects will be randomly assigned to receive either the test lens or the control lens in both eyes.

ELIGIBILITY:
Inclusion Criteria:

Note: All criteria apply to each eye

* Minimum 22 years of age
* Bilateral cataracts for which phacoemulsification extraction and posterior IOL implantation have been planned for both eyes
* Preoperative best corrected distance visual acuity (BCDVA) of 20/40 Snellen (0.5 Decimal) or worse with or without a glare source
* Potential for postoperative BCDVA of 20/30 Snellen (0.66 Decimal) or better
* Corneal astigmatism:

  * Normal corneal topography and no irregular corneal astigmatism
  * Preoperative corneal astigmatism of 2.50 D or less in both eyes, including posterior corneal astigmatism (PCA) and surgically induced astigmatism (SIA)
* Clear intraocular media, other than cataract
* Availability, willingness and sufficient cognitive awareness to comply with examination procedures
* Signed informed consent and HIPAA authorization or equivalent documentation necessary to comply with applicable privacy laws pertaining to medical treatment in the governing countries
* Ability to understand and respond to a questionnaire in English or the local language in which the informed consent and questionnaires are provided

Exclusion Criteria:

* Note: All criteria apply to each eye

  * Requiring an intraocular lens power outside the available range of +17.0 D to +26.0 D
  * Pupil abnormalities (non-reactive, fixed pupils, or abnormally shaped pupils)
  * Recent ocular trauma or ocular surgery that is not resolved/stable or may affect visual outcomes or increase risk to the subject
  * Prior corneal refractive (LASIK, LASEK, RK, PRK, etc.) or intraocular surgery
  * Corneal abnormalities such as stromal, epithelial or endothelial dystrophies that are predicted to cause visual acuity losses to a level of 20/30 Snellen (0.66 Decimal) or worse during the study
  * Inability to achieve keratometric stability for contact lens wearers (see Section 9.3)
  * Subjects with diagnosed degenerative visual disorders (e.g., macular degeneration or other retinal disorders) that are predicted to cause visual acuity losses to a level of 20/30 Snellen or worse during the study
  * Subjects with conditions associated with increased risk of zonular rupture, including capsular or zonular abnormalities that may lead to IOL decentration or tilt, such as pseudoexfoliation, trauma, or posterior capsule defects
  * Use of systemic or ocular medications that may affect vision Prior, current, or anticipated use during the course of the 6-month study of tamsulosin or silodosin (e.g., Flomax, Flomaxtra, Rapaflo) that may, in the opinion of the investigator, confound the outcome or increase the risk to the subject (e.g., poor dilation or a lack of adequate iris structure to perform standard cataract surgery)
  * Inability to focus or fixate for prolonged periods of time (e.g., due to strabismus, nystagmus, etc.)
  * Poorly-controlled diabetes
  * Acute, chronic, or uncontrolled systemic or ocular disease or illness that, in the opinion of the investigator, would increase the operative risk or confound the outcome(s) of the study (e.g., immunocompromised, connective tissue disease, suspected glaucoma, glaucomatous changes in the fundus or visual field, ocular inflammation, etc.). Note: controlled ocular hypertension without glaucomatous changes is acceptable.
  * Known ocular disease or pathology that may affect visual acuity or that may be expected to require retinal laser treatment or other surgical intervention during the course of the study (macular degeneration, cystoid macular edema, diabetic retinopathy, etc.)
  * Patient is pregnant, plans to become pregnant, is lactating or has another condition associated with the fluctuation of hormones that could lead to refractive changes
  * Concurrent participation or participation within 30 days prior to preoperative visit in any other clinical trial
  * Desire for monovision correction

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2025-01-01 (Estimated); Primary Completion 2025-07-01 (Estimated); Study Completion 2025-07-01 (Estimated)

PRIMARY OUTCOMES:
mean monocular, photopic BCDVA | 3 months postoperative

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Surgical Vision Clinical Trials, Study Director — Johnson & Johnson Surgical Vision

IPD SHARING:
Plan to Share IPD: Yes
Johnson & Johnson Medical Devices Companies have an agreement with the Yale Open Data Access (YODA) Project to serve as the independent review panel for evaluation of requests for clinical study reports and participant level data from investigators and physicians for scientific research that will advance medical knowledge and public health. Requests for access to the study data can be submitted through the YODA project site at http://yoda.yale.edu
URL: http://yoda.yale.edu